CLINICAL TRIAL: NCT05965167
Title: A Phase 1b, Open-label, Partially Randomised Study to Assess Safety and Compare Pharmacokinetics of New Oral hPTH(1-34) Tablet Formulations vs. Oral EBP05 Tablets and Subcutaneous Forteo® Injection in Healthy Male Subjects
Brief Title: Assess Safety and Compare PK of New Oral hPTH(1-34) Tablet Formulations vs. EBP05 Tablets and Subcutaneous Forteo
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENT-11-2023
Record Dates: First submitted 2023-06-08; First posted 2023-07-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hypoparathyroidism; Osteoporosis; Fractures, Bone; Other Disease
Keywords: Hypoparathyroidism; PTH(1-34); Parathyroid Hormone; Teriparatide; Osteoporosis
MeSH Terms: conditions — Hypoparathyroidism; Osteoporosis; Fractures, Bone; Disease | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Treatment A EBP05 2.5 mg (Experimental): Single dose of oral EBP05 2.5 mg
  Interventions: Drug: EBP05
- Treatment B EBP05 1.5 mg (Experimental): Single dose of oral EBP05 1.5 mg
  Interventions: Drug: EBP05
- Treatment C Forteo 0.02 mg (Experimental): Single SC injection of Forteo 0.02 mg
  Interventions: Drug: Forteo 0.02 mg
- Treatment D EBP11 1.5 mg (Experimental): Single dose of oral EBP11 1.5 mg
  Interventions: Drug: EBP11
- Treatment E EBP11 BID (dose determined after IA) (Experimental): BID administration of oral EBP11 2.5 mg tablets
  Interventions: Drug: EBP11
- Treatment F EBP11 BID (dose determined after IA) (Experimental): BID administration of oral EBP11 tablets 1.5 mg tablets (3 x 0.5 mg tablets) as first dose and 2.5 mg (5 x 0.5 mg tablets) as second dose.
  Interventions: Drug: EBP11
- Treatment G EBP11 1.5 mg (Experimental): Single dose of oral EBP11 1.5 mg
  Interventions: Drug: EBP11
- Treatment I EBP22 1.5 mg (Experimental): Single dose of oral EBP22 1.5 mg
  Interventions: Drug: EBP22
- Treatment J EBP22 1.5 mg (Experimental): Single dose of oral EBP22 1.5 mg
  Interventions: Drug: EBP22
- Treatment K EBP05 1.5 mg (Experimental): Single dose of oral EBP05 1.5 mg
  Interventions: Drug: EBP05
- Treatment L EBP05 2.5 mg (Experimental): Single dose of oral EBP05 2.5 mg
  Interventions: Drug: EBP05
- Treatment M Forteo 0.02 mg (Experimental): Single SC injection of Forteo 0.02 mg
  Interventions: Drug: Forteo 0.02 mg
- Treatment N EBP05 3.0 mg (Experimental): Single dose of oral EBP05 3.0 mg
  Interventions: Drug: EBP05
- Treatment H EBP22 2.5 mg (5 x 0.5 mg). (Experimental): Single dose of oral EBP22 2.5 mg (5 x 0.5 mg).
  Interventions: Drug: EBP22
- Treatment O EBP05 2.5 mg (Experimental): Single dose of oral EBP05 2.5 mg
  Interventions: Drug: EBP05
- Treatment P EBP11-F2 1.5 mg (Experimental): Single dose of oral EBP11-F2 1.5 mg
  Interventions: Drug: EBP11-F2
- Treatment Q EBP11-F4 2.5 mg (Experimental): Single dose of oral EBP11-F4 2.5 mg
  Interventions: Drug: EBP11-F4
- Treatment R EBP05 2.5 mg (Experimental): Single dose of oral EBP05 2.5 mg
  Interventions: Drug: EBP05
- Treatment S EBP05 2.5 mg (Experimental): Single dose of oral EBP05 2.5 mg
  Interventions: Drug: EBP05

INTERVENTIONS:
Drug: EBP05 — Oral tablets
  Other Names: hPTH(1-34)
  Arms: Treatment A EBP05 2.5 mg; Treatment B EBP05 1.5 mg; Treatment K EBP05 1.5 mg; Treatment L EBP05 2.5 mg; Treatment N EBP05 3.0 mg; Treatment O EBP05 2.5 mg; Treatment R EBP05 2.5 mg; Treatment S EBP05 2.5 mg
Drug: Forteo 0.02 mg — Subcutaneous injection
  Other Names: hPTH(1-34)
  Arms: Treatment C Forteo 0.02 mg; Treatment M Forteo 0.02 mg
Drug: EBP11 — Oral tablets
  Other Names: hPTH(1-34)
  Arms: Treatment D EBP11 1.5 mg; Treatment E EBP11 BID (dose determined after IA); Treatment F EBP11 BID (dose determined after IA); Treatment G EBP11 1.5 mg
Drug: EBP22 — Oral tablets
  Other Names: hPTH(1-34)
  Arms: Treatment H EBP22 2.5 mg (5 x 0.5 mg).; Treatment I EBP22 1.5 mg; Treatment J EBP22 1.5 mg
Drug: EBP11-F2 — Oral tablets
  Other Names: hPTH(1-34)
  Arms: Treatment P EBP11-F2 1.5 mg
Drug: EBP11-F4 — Oral tablets
  Other Names: hPTH(1-34)
  Arms: Treatment Q EBP11-F4 2.5 mg

SUMMARY:
The purpose of this study is to characterize and compare the pharmacokinetics of hPTH(1 34) after treatment with modified oral formulations (EBP11, EBP11-F2, EBP11-F4 and EBP22) versus three dose levels of Entera Bio's extensively studied oral EBP05 1.5 mg, 2.5 mg and 3.0 mg as well as the commercial Forteo 0.02 mg subcutaneous injection.

DETAILED DESCRIPTION:
Stated in summary, eligibility criteria and outcome measures

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18 - 35 years of age, inclusive, at screening.
2. Continuous nonsmoker who has not used nicotine containing products (including e-cigarettes, vapors, etc.) for at least 12 months prior to first dosing and throughout the study, based on subject self-reporting.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical condition, physical examination, laboratory profiles, vital signs, orthostatic vital sign measurements, or ECGs, as deemed by the PI or designee to be relevant to the study and does not pose an additional risk to the subject by their participation in the study.
5. Understands the study procedures described in the Informed Consent Form (ICF), be willing and able to comply with the protocol, and provides written consent.

Exclusion Criteria:

1. History or current condition of mental instability or cognitive impairment that, in the opinion of the investigator, could compromise the validity of informed consent, compromise the safety of the participant, or lead to nonadherence with the study protocol or inability to conduct the study procedures.
2. Active gastrointestinal inflammatory disorder, gastrointestinal motility disorders, and chronic gastritis, including but not limited to: ulcerative colitis, Crohn's disease, irritable bowel syndrome, short bowel syndrome, celiac disease, gastroparesis, that may affect drug bioavailability.
3. Any conditions or factors that, in the judgment of the PI or designee, somehow may impact gastrointestinal absorption, distribution or metabolism of parathyroid hormone analogues, or known to potentiate or predispose to undesired effects.
4. History of significant gastrointestinal, liver or kidney disease, or gastrointestinal surgery (including bariatric surgery, or any other interventional procedures with stomach and intestinal tract) that may affect either drug bioavailability, or hPTH(1-34) or SNAC metabolism.
5. History or presence of alcohol or drug abuse or positive urine drug or blood alcohol results at screening.
6. Known allergies or sensitivities to components of the Study Medication (e.g. soy) or known hypersensitivity to PTH or hPTH(1-34).
7. History or presence of clinically significant:

   * Urolithiasis;
   * Angina at Screening, in the opinion of the PI;
   * Hypocalcemia or hypercalcemia at screening;
   * Personal or family history of congenital long QT syndrome or known family history of sudden death.
8. Subjects with ECG findings deemed abnormal with clinical significance by the PI or designee at screening for the following:

   * QTcF interval > 470 msec;
   * PR > 220 msec;
   * QRS > 120 msec.
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
10. Seated blood pressure is less than 90 systolic or 40 diastolic mmHg or greater than 140 systolic or 90 diastolic mmHg at screening;
11. Orthostatic vital sign results with a decrease in systolic > 20 mmHg or decrease in diastolic > 10 mm Hg, and/or increase in heart rate of > 20 beats per minute at screening or Day 1 check-in.
12. Seated heart rate is lower than 50 bpm or higher than 99 bpm at screening (when clinically significant as determined by PI).
13. Estimated creatinine clearance < 80 mL/min at screening
14. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and nonprescription medications, herbal remedies, or vitamin supplements that should be taken on the treatment visit day before the dosing of Study Medication and 2 hours after the dosing of Study Medication.
    * H2 blocker or PPI or antacid (including prescription and nonprescription) three days before the dosing of the Study Medication and 2 hours after the dosing of Study Medication.
15. Donation of blood or significant blood loss within 56 days prior to first dosing.
16. Hemoglobin levels below 13 g/dL at screening or at in screening test done during the study.
17. Plasma donation within 7 days prior to first dosing.
18. Participation in another interventional clinical study within 30 days prior to screening visit.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the pharmacokinetic profile of plasma hPTH(1-34) after single or twice daily oral administration for treatment regimen as listed under Arms and Interventions at 5, 10, 15, 20, 40, 50, 60, 75, 90, 105, 120, 180, 240, 360 min. post dose | 6 hours
  Pharmacokinetic parameter - plasma hPTH(1-34) in pg/mL
Calculation of plasma levels of hPTH(1-34) AUC0-t for each treatment regimen | 6 hours
  Pharmacokinetic parameter - total drug exposure at different time points up to 360 min. post dose
Calculation of plasma levels of hPTH(1-34) AUC0-inf for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - total drug exposure in pg/mL over time from 0 extrapolated to infinity
Calculation of plasma levels of hPTH(1-34) AUC%extrap for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - Percent of AUC0-inf extrapolated to confirm reliability
Calculation of plasma levels of hPTH(1-34) Cmax for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - hPTH (1-34) maximal concentration in pg/mL (Cmax)
Calculation of plasma levels of hPTH(1-34) Tmax for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - time in minutes to reach max. concentration of hPTH(1-34)
Calculation of plasma levels of hPTH(1-34) Kel for each treatment regimen | 6 hours
  Pharmacokinetic parameter - elimination rate constant in pg/mL, fraction of drug eliminated per time-point up to 360 min. post dose
Calculation of plasma levels of hPTH(1-34) t½ for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - terminal elimination half life of hPTH(1-34) in minutes
Calculation of plasma levels of hPTH(1-34) Tlast for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - time of the last measurable concentration of hPTH(1-34) in minutes
Assessment of inter-subject variability of hPTH(1-34) for each treatment regimen | 6-14 hours
  Pharmacokinetic parameter - Coefficient of Variance (CV%) of hPTH (1-34)
Calculation of dose proportionality for hPTH(1-34) for relevant treatment regimen | 6 hours
  Pharmacokinetic parameter
Assessment of the duration of exposure to hPTH(1-34) in minutes | 6 hours
  Pharmacokinetic parameter - up to 360 min. post dose
Vital Signs - body temperature (Celsius) | 6 hours
  Safety parameter (group mean at each time point up to 360 min. post dose)
Vital Signs - respiratory rate (breaths per minute) | 6 hours
  Safety parameter (group mean at each time point up to 360 min. post dose)
Vital Signs - blood pressure (systolic/diastolic mmHg) | 6 hours
  Safety parameter (group mean at each time point up to 360 min. post dose)
Vital Signs - heart rate (beats per minute) | 6 hours
  Safety parameter (group mean at each time point up to 360 min. post dose)
Incidence of Treatment-Emergent Adverse Events as assessed by the Principle Investigator | 6-14 hours
  Safety parameter - AEs observed over duration of study participation
Incidence of Serious Adverse Events (SAEs) as assessed by the Principle Investigator | 6-14 hours
  Safety parameter - SAEs observed over duration of study participation

OTHER OUTCOMES:
Measurement of plasma soybean trypsin inhibitor, Kunitz type (SBTI) levels (EBP05 only) | 6 hours
  Pharmacokinetic parameter in ng/mL
Measurement of plasma salcaprozate sodium (SNAC) levels (EBP05 only) | 6 hours
  Pharmacokinetic parameter in μg/mL
Measurement of serum calcium (albumin-corrected total calcium) for all treatment regimen | 6 hours
  Pharmacodynamic parameter in mg/dL at 120, 240, 360 min post dose
Measurement of serum phosphate for all treatment regimen | 6 hours
  Pharmacodynamic parameter in mg/dL at 120, 240, 360 min post dose
Measurement of serum intact hPTH(1-84) for all treatment regimen | 6 hours
  Pharmacodynamic parameter in pg/mL at 120, 240, 360 min post dose
Measurement of serum 1,25-(OH)2D for all treatment regimen (optional) | 6 hours
  Pharmacodynamic parameter in ng/mL at 120, 240, 360 min post dose
Assessment of food effect on EBP05 PK profile | 60 minutes
  Pharmacokinetic parameter measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Caraco, MD, Principal Investigator — Clinical Research Center Hadassah Ein Kerem Medical Center
Locations (1):
- Clinical Research Center Hadassah Ein Kerem Medical Center, Jerusalem, Israel